CLINICAL TRIAL: NCT07181213
Title: Genetic Predisposition to High Blood Pressure
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Oliver Gimm, Professor of Surgery, Linkoeping University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: Dnr 2024-07874-01
Record Dates: First submitted 2025-09-12; First posted 2025-09-18 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Hypertension; Primary Aldosteronism; Genetic Predisposition to Disease
MeSH Terms: conditions — Hypertension; Hyperaldosteronism; Genetic Predisposition to Disease | interventions — Adrenalectomy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Presence of unilateral primary aldosteronism in patients with genetic variant and hypertension (Active Comparator): Unilateral adrenalectomy is offered
  Interventions: Procedure: Adrenalectomy
- Presence of bilateral primary aldosteronism in patients with genetic variant and hypertension (No Intervention): Medical treatment is offered

INTERVENTIONS:
Procedure: Adrenalectomy — Surgical removal of patients with unilateral primary aldosteronism in patients selected by the presence of a genetic variant and hypertension
  Arms: Presence of unilateral primary aldosteronism in patients with genetic variant and hypertension

SUMMARY:
Primary aldosteronism (PA) is a known but underdiagnosed cause of high blood pressure. It is estimated that more than 10% of all people with high blood pressure (HT) suffer from PA, which is often caused by aldosterone-producing adrenal cortical tumors (APAs).

In a pilot study with 35 patients with APAs leading to hypertension, the investigators have identified a genetic variant in a presumed Calcium-channel gene. The variant was significantly overrepresented in patients with APAs compared to the normal population (12% compared to approximately 4%). Interestingly, all patients having APAs and the variant were men.

The SCAPIS study is a world-unique Swedish research study in the field of heart/lungs, in which 30,000 randomly selected people between the ages of 50-64 participated. The study is a collaboration between the universities of Gothenburg, Lund, Linköping, Uppsala and Umeå, as well as the Karolinska Institute in Stockholm. In Linköping, about 5,000 persons participated.

The investigators have now screened 4762 persons from the SCAPIS study for this variant and found it in little less than 6%. Overall, patients with the variant had more often been diagnosed with HT and were mote often treated for HT as well. Interestingly, this difference was only found in men.

The investigators now want to investigate the following:

1. identify those persons with the genetic variant and HT that have PA,
2. identify those persons with PA that have APAs/unilateral disease,
3. identify how many patients with APAs/unilateral disease can be cured by surgery.

ELIGIBILITY:
Inclusion Criteria:

* patients that participated in the SCAPIS study
* patients that have a particular genetic variant
* patients that have hypertension

Exclusion Criteria:

* patients who do not want to participate
* patients who cannot give consent
* patients who are too sick to be operated

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2026-01-01 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Normal aldosterone-renin-ratio | 6 months following surgery

SECONDARY OUTCOMES:
Blood pressure both systolic and diastolic | 6 months after surgery
Number of antihypertensive drugs | 6 months following surgery
Normal potassium level | 6 months postoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- Linköping University Hospital, Linköping, Östergötland County, Sweden

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication